CLINICAL TRIAL: NCT00912431
Title: A Pharmacokinetic and Exploratory Biomarker Study of ABT-126 in the Cerebrospinal Fluid (CSF) of Healthy Subjects
Brief Title: Pharmacokinetic and Exploratory Biomarker Study of ABT-126 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Daniel Llano, MD, PhD/Associate Medical Director, Abbott
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: M11-061
Record Dates: First submitted 2009-06-02; First posted 2009-06-03 (Estimated); Last update posted 2010-11-02 (Estimated); Status verified 2010-09

CONDITIONS: Healthy
Keywords: Healthy Volunteers
MeSH Terms: interventions — ABT-126

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: ABT-126
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ABT-126 — ABT-126 administered on Day 1 of Period 1
  Arms: 1
Drug: Placebo — Placebo for ABT-126 administered on Day 1 of Period 2
  Arms: 2

SUMMARY:
The objectives of this study are to determine the cerebrospinal fluid (CSF) levels of ABT-126 and to examine the effects of ABT-126 on exploratory biomarkers after administration of a single does of ABT-126 in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects between 18 and 50 years of age

Exclusion Criteria:

* History of bleeding disorders or Deep Vein Thrombosis
* History of spinal surgery
* History of migraine headaches, or other types of headaches occuring more than 2 times per month, or history of spinal disc disease, or chronic, significant low back pain

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2009-06; Primary Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability Assessments (i.e., ECG, clinical laboratory tests, vital signs, weight, AE assessment, physical examination and neurological examination) | Day 1 thru Day 4 in Periods 1 and 2
Pharmacokinetic samples | Day 1 (up to 24-hour post dose) in Periods 1 and 2
Cerebrospinal Fluid samples | Day 1 (up to 24-hour post dose) in Periods 1 and 2

CONTACTS AND LOCATIONS:
Locations (1):
- Site Reference ID/Investigator# 20761, Glendale, California, United States